

Title: Special drug use surveillance of Takecab tablets for "prevention of recurrence of gastric/duodenal ulcer in patients receiving low-dose aspirin:long-term use"

NCT Number: NCT03214094

Statistical analysis plan Approve Date: 07-AUG-2019

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

(Analysis of final results)

| Takecab | <b>Tablets</b> |
|---------|----------------|
| | Takecab |

Title of Surveillance : Prevention of recurrent gastric or duodenal ulcer during low-dose

aspirin therapy: long-term use

Protocol No. : Vonoprazan-5004

Sponsor : Takeda Pharmaceutical Company Limited

| PPD | |
|-----|---------|
| PPD | |
| | PPD<br> |
| PPD | |

# Table of contents

| L | ist of ter | ms/abbreviations | 3 |
|---|---|---|---|
| A | nalysis s | et | 5 |
| In | nportant | identified risks, important potential risks, and important missing information | 6 |
| Н | andling | of TIME WINDOW | 8 |
| Η | andling | of others | 9 |
| 1 | Numbe | er of medical institutions, number of patients enrolled, and patient disposition | 10 |
| | 1.1 Bı | reakdown of patients (figure of patient disposition) | 10 |
| 2 | Patient | demographics | 12 |
| | 2.1 Pa | tient demographics | 12 |
| 3 | Treatm | ent details and concomitant drug | 14 |
| | 3.1 St | atus of treatment with Takecab Tablets | 14 |
| | 3.2 St | atus of low-dose aspirin therapy | 14 |
| | 3.3 Co | oncomitant drug (excluding low-dose aspirin) | 14 |
| 4 | Tabula | ted analysis on safety results | 16 |
| | 4.1 In | cidence of AE and ADR/infection | 16 |
| | 4.1.1 | Incidence of AE | 16 |
| | 4.1.2 | Incidence of ADR/infection | 17 |
| | 4.1.3 | Incidence of AE and ADR/infection falling under the categories of important | |
| | | identified risks, important potential risks, and important missing information | 18 |
| | 4.2 In | cidence of AE and ADR/infection in patients excluded from safety evaluation | 19 |
| | 4.2.1 | Incidence of AE | 19 |
| | 4.2.2 | Incidence of ADR/infection | 20 |
| | 4.3 In | cidence of AE and ADR/infection by seriousness, time of onset, and outcome | 21 |
| | 4.3.1 | Incidence of AE by seriousness, time of onset, and outcome | 21 |
| | 4.3.2 | Incidence of ADR/infection by seriousness, time of onset, and outcome | 22 |
| | 4.4 In | cidence of ADR/infection by factor of patient demographics and treatment details | 23 |
| | 4.4.1 | Incidence of ADR/infection by factor of patient demographics and treatment details. | 23 |
| | 4.4.2 | Incidence of ADR/infection by sex | 24 |
| | 4.4.3 | Incidence of ADR/infection by age subgroup | 25 |
| | 4.4.4 | Incidence of ADR/infection by purpose of low-dose aspirin therapy | 25 |
| | 4.4.5 | Incidence of ADR/infection by presence/absence of complication | 26 |
| | 4.4.6 | Incidence of ADR/infection by presence/absence of renal disease | 26 |
| | 4.4.7 | Incidence of ADR/infection by presence/absence of hepatic disease | 26 |
| | 4.4.8 | Incidence of ADR/infection by BMI subgroup | 27 |
| | 4.4.9 | Incidence of ADR/infection by initial daily dose of low-dose aspirin | 27 |

| | 4.4.10 Incidence of ADR/infection by presence/absence of concomitant drug (exclu | ding |
|---|---|---|
| | low-dose aspirin) | 28 |
| | 4.4.11 Change of liver function test value | 28 |
| 5 | Tabulated analysis on efficacy results | 29 |
| | 5.1 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach | or |
| | duodenum | 29 |
| | 5.2 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach | or |
| | duodenum (count in each subgroup) | 29 |
| 6 | Incidence of ADR/infection in additional pharmacovigilance activities | 31 |
| | 6.1 Incidence of ADR/infection in additional pharmacovigilance activities (Attachme | nt |
| | Form 12) | 31 |
| 7 | Outline of patients in postmarketing surveillance, etc | 32 |
| | 7.1 Outline of patients in postmarketing surveillance, etc. (Attachment Form 16) | 32 |
| R | Revision history (version control) | 33 |

#### List of terms/abbreviations

- The drug: Takecab Tablets
- ADR, etc.: Abbreviation of "adverse reaction and infection". Adverse events other than those which the surveillance investigator assessed the causality as "not related". In this statistical analysis plan, the term "ADR/infection" is used in the title, and the term "ADR, etc." is used in the text and tables.
- Serious adverse event:
  - An adverse event which the surveillance investigator assessed as "serious". Events included
    in the MedDRA code list of Takeda Medially Significant AE List are handled as serious
    even if the surveillance investigator assessed as "non-serious".
- Causality "related" to Takecab Tablets: The causality of an event not assessed as "not related" to Takecab Tablets is handled as "related", and the causality of an event assessed as "not related" to Takecab Tablets is handled as "not related".
- Summary statistics: An inclusive term of number of patients, mean, standard deviation, maximum value, minimum value, and quartile.
- Treatment days: The day before Takecab Tablets is started is Day -1, and the day when Takecab Tablets is started is Day 1.
- Duration (days) of treatment with Takecab Tablets: Completion date of treatment with Takecab
   Tablets start date of treatment with Takecab Tablets + 1 (excluding days without treatment)
  - For patients with "under treatment with Takecab Tablets 12 months after the start of treatment" entered on the survey form, the duration of treatment is handled as 365 days (excluding days without treatment).
- Duration (days) of low-dose aspirin therapy: Completion date of low-dose aspirin therapy start date of low-dose aspirin therapy + 1 (excluding days without treatment)
  - For patients with missing completion date of low-dose aspirin therapy or "under low-dose
    aspirin therapy at the completion of survey" entered on the survey form, the duration of
    therapy is handled as missing (unknown).
  - For other patients with "therapy started before the start of treatment with Takecab Tablets" described as the status of low-dose aspirin on the survey form, but with missing start date, the duration of therapy is calculated by imputing "start time of low-dose aspirin therapy" described as patient demographics (the first date of the month is the start date of therapy). If only the month is missing, "January 1" is imputed as the start date of therapy. Otherwise

(both the year and month are missing or "unknown"), the duration of therapy is handled as missing (unknown).

- Patients whose survey forms have not been collected: In patients enrolled in the survey, patients
  whose survey forms have not been collected.
- Patients whose survey forms have been collected: In patients enrolled in this survey, patients
  whose survey forms have been collected.
- BMI (kg/m²): Calculated as Weight (kg)/Height (m)² (rounded to the first decimal place).
- Time of onset of AE (or ADR, etc.): When onset date of an AE (or ADR, etc.) is unknown, the first date of the month is the onset date. However, when the year and month of the start of Takecab Tablets and the year and month of AE (or ADR, etc.) onset are the same, the time of onset is allocated as the first start date of Takecab Tablets.

#### Analysis set

In this survey, two analysis sets of "safety analysis set" and "efficacy analysis set" will be set. Individual analysis sets are defined as below.

# Safety analysis set

In this statistical analysis plan, "safety analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for safety". In the patients whose survey forms have been collected, those falling under the following categories are excluded from the safety analysis set.

- Takecab Tablets was not administered
- Administration of Takecab Tablets prior to contract period [found later]
- Enrollment in this survey 15 days or later after prescription of Takecab Tablets [found later]
- It is unknown whether any AE developed or not

### Efficacy analysis set

In this statistical analysis plan, "efficacy analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for efficacy". In the safety analysis set, patients falling under the following categories are excluded from the efficacy analysis set.

- Other than target disease [found later]
- Patient failing to meet all of the inclusion criteria
- Patient meeting any of the exclusion criteria
- Patient with no post-baseline efficacy data
  - A post-baseline examination was not conducted or was conducted outside the time window to determine the "development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum."

### Important identified risks, important potential risks, and important missing information

- Important identified risk: Not applicable
- Important potential risk
  - Hepatic function disorder: An AE falling under SMQ code 20000006 (Drug related hepatic disorders - comprehensive search [SMQ] narrow) is handled as hepatic function disorder.
  - Fracture: An AE falling under any of the PT codes listed in Table 1 is handled as fracture.
  - Gastrointestinal infection with clostridium difficile: An AE falling under SMQ code 20000080 (Pseudomembranous colitis [SMQ] narrow) is handled as gastrointestinal infection with clostridium difficile.
  - Neuroendocrine tumour due to increased serum gastrin: An AE falling under SMQ code 20000090 (Malignancies [SMQ] narrow) is handled as neuroendocrine tumour due to increased serum gastrin.
- Important missing information: Not applicable

Table 1 Fracture-related PT codes

| PT NAME | PT CODE | PT NAME | PT CODE |
|---|---|---|---|
| Acetabulum fracture | 10000397 | Ilium fracture | 10021343 |
| Ankle fracture | 10002544 | Impacted fracture | 10066386 |
| Atypical femur fracture | 10070884 | Jaw fracture | 10023149 |
| Atypical fracture | 10072395 | Limb fracture | 10074551 |
| Avulsion fracture | 10066184 | Lower limb fracture | 10061599 |
| Bone fissure | 10064210 | Lumbar vertebral fracture | 10049947 |
| Bone fragmentation | 10064211 | Maisonneuve fracture | 10081343 |
| Cervical vertebral fracture | 10049946 | Metaphyseal corner fracture | 10079667 |
| Chance fracture | 10073162 | Multiple fractures | 10028200 |
| Clavicle fracture | 10009245 | Open fracture | 10030527 |
| Comminuted fracture | 10052614 | Osteophyte fracture | 10080550 |
| Complicated fracture | 10010149 | Osteoporotic fracture | 10031290 |
| Compression fracture | 10010214 | Patella fracture | 10034122 |
| Craniofacial fracture | 10077603 | Pathological fracture | 10034156 |
| Cuboid syndrome | 10081921 | Pelvic fracture | 10061161 |
| Epiphyseal fracture | 10053962 | Pubis fracture | 10070286 |

| PT NAME | PT CODE | PT NAME | PT CODE |
|---|---|---|---|
| Facial bones fracture | 10016042 | Radius fracture | 10037802 |
| Femoral neck fracture | 10016450 | Rib fracture | 10039117 |
| Femur fracture | 10016454 | Sacroiliac fracture | 10074362 |
| Fibula fracture | 10016667 | Scapula fracture | 10039579 |
| Foot fracture | 10016970 | Skull fracture | 10061365 |
| Forearm fracture | 10016997 | Skull fractured base | 10040960 |
| Fracture | 10017076 | Spinal compression fracture | 10041541 |
| Fracture blisters | 10079423 | Spinal fracture | 10041569 |
| Fracture displacement | 10053206 | Spinal fusion fracture | 10074807 |
| Fracture malunion | 10017085 | Stapes fracture | 10081442 |
| Fracture nonunion | 10017088 | Sternal fracture | 10042015 |
| Fracture of clavicle due to birth trauma | 10017107 | Stress fracture | 10042212 |
| Fractured coccyx | 10049164 | Subchondral insufficiency fracture | 10079864 |
| Fractured ischium | 10017290 | Thoracic vertebral fracture | 10049948 |
| Fractured sacrum | 10017308 | Tibia fracture | 10043827 |
| Fractured skull depressed | 10017310 | Torus fracture | 10066094 |
| Greenstick fracture | 10018720 | Traumatic fracture | 10049514 |
| Hand fracture | 10019114 | Ulna fracture | 10045375 |
| Hip fracture | 10020100 | Upper limb fracture | 10061394 |
| Humerus fracture | 10020462 | Wrist fracture | 10048049 |

# **Handling of TIME WINDOW**

Data of tests/observations/endpoints which are evaluable (i.e., data which are not missing and are considered to be adopted) are handled based on the following details.

Data which are evaluable and within the time window will be adopted. If there are multiple evaluable data within the same time window, the nearest date of test/observation/assessment to the standard day will be adopted. If the number of days from the standard day is the same or the standard day is not specified, data of the later date will be adopted. The difference from the standard day is determined based on the post-treatment days.

Laboratory tests (AST, ALT, γ-GTP, ALP, Total bilirubin, LDH, Serum gastrin)

| Assessment time | Standard day of conduct | Time window Post-treatment days |
|---|---|---|
| At the start of treatment | Post-treatment days: -1 | -8 to 1 |
| At the completion of survey | Post-treatment days: – | 2 or more |

Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum

| Assessment time | Standard day of conduct | Time window Post-treatment days |
|---|---|---|
| At the completion of survey | Post-treatment days: – | 2 or more |

# Handling of others

• None particularly

#### 1 Number of medical institutions, number of patients enrolled, and patient disposition

### 1.1 Breakdown of patients (figure of patient disposition)

Analysis All patients enrolled in this survey (patients enrolled)

population:

Analysis items: Patients enrolled

Number of medical institutions

Patients whose survey forms have not

been collected

Patients whose survey forms have been

collected

Patients excluded from safety

evaluation\*

Reason of exclusion (multiple

counts)

[Takecab Tablets not administered,

Administration prior to contract

period [found later], Enrollment 15 days or later after prescription of Takecab Tablets [found later], Unknown whether any AE

developed or not]

Patients targeted for safety evaluation\*

Patients excluded from efficacy

evaluation\*

Reason of exclusion (multiple

counts)

[Other than target disease [found later],

Patient failing to meet all of the inclusion criteria, Patient meeting any of the exclusion criteria, Patient with no post-baseline efficacy data

Patients targeted for efficacy

evaluation\*

Analysis method:

Following analysis will be conducted for the above analysis items, and a figure of patient disposition will be prepared.

The number of medical institutions will also be calculated concerning patients enrolled in the survey. If patients are enrolled in more than one department in one medical institution, the number of the medical institution is counted as one. Number of patients excluded from safety evaluation and efficacy evaluation are counted by reason of exclusion, and a list will be prepared.

- \* "Patients targeted for safety evaluation" indicates "safety analysis set".

  "Patients excluded from safety evaluation" indicates patients excluded from

  "safety analysis set". "Patients targeted for efficacy evaluation" indicates

  "efficacy analysis set". "Patients excluded from efficacy evaluation" indicates

  patients excluded from "efficacy analysis set" in "safety analysis set".
- (1) Frequency count

#### 2 Patient demographics

#### 2.1 Patient demographics

Analysis Safety analysis set

population:

Analysis items: Sex [Male, Female]

Age (year)  $[Min \le -.. < 65, \ge 65 \le -.. < 75, \ge 75 \le -.. \le Max]$ 

Previous medical history [Gastric ulcer, Duodenal ulcer]

(multiple counts)

Purpose of low-dose aspirin [Angina pectoris, Myocardial infarction,

therapy (multiple counts)

Transient ischemic attack (TIA), Cerebral

infarction, Others]

Existence of coronary arterial [Yes or No]

stent

Inpatient/outpatient [Outpatient, Inpatient]

classification

Existence of hypersensitivity [Yes or No or Unknown]

predisposition

Existence of complication [Yes or No]

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$  [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le - \le Max$ 

Existence of *H. pylori* infection [Positive or Negative or Unknown]

Smoking history [Non-smoker, Current smoker, Ex-smoker,

Unknown]

Drinking history [Yes or No or Unknown]

Existence of stress, a risk factor [Yes or No or Unknown]

for developing gastric or

duodenal ulcer

Existence of acid-suppressant [Yes or No or Unknown]

therapy before the start of

treatment with Takecab Tablets

to prevent recurrent gastric or

duodenal ulcer

Breakdown of drugs in patients [Lansoprazole, Omeprazole, Rabeprazole,

with "Yes" Esomeprazole, H<sub>2</sub>-blocker]

Analysis method: Following analysis will be conducted for the above analysis items.

| (1) Frequency counts of countable data, and summary statistics of quantitative data |
|---|

### 3 Treatment details and concomitant drug

#### 3.1 Status of treatment with Takecab Tablets

Analysis Safety analysis set

population:

Analysis items: Initial daily dose of Takecab [10 mg, Others]

Tablets

Duration (days) of treatment [1<= - <=84, 85<= - <=168, 169<= - <=Max]

with Takecab Tablets

Reasons for discontinuation [Incidence of AE, No patient visit due to reasons

of treatment with Takecab such as changing hospital, Pregnancy,

Tablets Development of gastric ulcer/duodenal

ulcer/hemorrhagic lesions in stomach or duodenum, Discontinuation of low-dose

aspirin therapy, Others]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative

data

# 3.2 Status of low-dose aspirin therapy

Analysis Safety analysis set

population:

Analysis items: Initial daily dose of low-dose [81 mg, 100 mg, 162 mg, 200 mg, Others]

aspirin

Duration (days) of low-dose [1<= - <=84, 85<= - <=168, 169<= - <=Max,

aspirin therapy Unknown]

Purpose of treatment with [Treatment of complication, Development of Takecah Tablets after the gastric ulcer/duodenal ulcer/hemorrhagic

Takecab Tablets after the gastric ulcer/duodenal ulcer/hemorrhagic completion of low-dose lesions in stomach or duodenum, Development

aspirin therapy of new gastrointestinal disease not mentioned above after treatment with Takecab Tablets,

Others (e.g., prophylactic treatment)]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative

data

#### 3.3 Concomitant drug (excluding low-dose aspirin)

Analysis Safety analysis set

population:

Analysis items: Existence of concomitant drug (excluding [Yes or No]

low-dose aspirin)

Type of concomitant drug (excluding low-dose aspirin)

Analysis method:

Following analysis will be conducted for the above analysis items. Concomitant drugs will be coded to terms in prescription drug term data file, and the data will be summarized by generic name. The drugs will be listed in descending order of frequency. When an identical drug (in generic name) is administered multiple times in one patient, one patient is counted for the drug (in generic name). When data of a generic name is missing, the product name will be applied.

(1) Frequency count

#### 4 Tabulated analysis on safety results

#### 4.1 Incidence of AE and ADR/infection

#### 4.1.1 Incidence of AE

Analysis Safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

 Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.1.2 Incidence of ADR/infection

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

# 4.1.3 Incidence of AE and ADR/infection falling under the categories of important identified risks, important potential risks, and important missing information

## 4.1.3.1 Incidence of AEs falling under the category of safety specification (count by risk)

Analysis Safety analysis set

population:

Analysis items: AEs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness

[Serious, Non-serious]

Analysis method: Following analyses will be conducted for the above analysis items in each

subgroup by risk. The risks are important identified risks, important potential

risks, and as defined in important missing information.

[Classification of AE]

 AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).

- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC. However, when the multiple events differ in
  seriousness, one patient will be counted as both serious and non-serious.
- PT will be presented with number and proportion of patients with AEs in
  ascending order of PT codes. When multiple events coded to terms in an
  identical PT developed in a single patient, one patient will be counted for
  the PT. However, when the multiple events differ in seriousness, one patient
  will be counted as both serious and non-serious.

# 4.1.3.2 Incidence ADRs/infections falling under the category of safety specification (count by risk)

Analysis Safety analysis set

population:

Analysis items: ADRs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness [Serious, Non-serious]

Analysis method: Following analyses will be conducted for the above analysis items in each subgroup by risk. The risks are important identified risks, important potential risks, and as defined in important missing information.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, when the multiple events differ in seriousness, one patient will be counted as both serious and non-serious.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, when the multiple events differ in seriousness, one patient will be counted as both serious and non-serious.

#### 4.2 Incidence of AE and ADR/infection in patients excluded from safety evaluation

#### 4.2.1 Incidence of AE

Analysis Patients excluded from safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- Number of patients with AEs (1)
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

Number of patients who experienced AEs.

[Number of incidence of AEs]

Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.2.2 Incidence of ADR/infection

Analysis Patients excluded from safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

 Number of ADRs, etc. which developed. When an ADR, etc. developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

 ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).

- SOC will be presented with number and proportion of patients with ADR,
   etc. in the internationally agreed order of SOC. When multiple events coded
   to terms in an identical SOC developed in a single patient, one patient will
   be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

### 4.3 Incidence of AE and ADR/infection by seriousness, time of onset, and outcome

#### 4.3.1 Incidence of AE by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: Adverse event

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset (days) [1<= - <=84, 85<= - <=168, 169<= - <=Max, Unknown]

Outcome [Resolved, Resolved, Resolved with

sequelae, Death (due to the relevant event), Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC. However, in an identical SOC, one event is adopted
  according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after Takecab Tablets was started

Outcome: Death (due to the relevant event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not resolved  $\rightarrow$  Resolving  $\rightarrow$  Resolved  $\rightarrow$  Unknown

#### 4.3.2 Incidence of ADR/infection by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset (days)  $[1 \le - \le 84, 85 \le - \le 168, 169 \le - \le Max,$ 

Unknown]

Outcome [Resolved, Resolving, Not resolved, Resolved with

sequelae, Death (due to the relevant event),

Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after Takecab Tablets was started

Outcome: Death (due to the relevant event)  $\rightarrow$  Resolved with sequelae  $\rightarrow$  Not resolved  $\rightarrow$  Resolving  $\rightarrow$  Resolved  $\rightarrow$  Unknown

# 4.4 Incidence of ADR/infection by factor of patient demographics and treatment details

### 4.4.1 Incidence of ADR/infection by factor of patient demographics and treatment details

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Age (year)  $[Min \le -.. \le 65, 65 \le -.. \le 75,$ 

 $75 \le - \le Max$ 

Purpose of low-dose aspirin therapy [Angina pectoris, Myocardial

(multiple counts) infarction, Transient ischemic attack

(TIA), Cerebral infarction, Others]

Existence of complication [Yes or No]
Existence of renal disease [Yes or No]
Existence of hepatic disease [Yes or No]

BMI  $(kg/m^2)$  [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le - \le Max$ 

Initial daily dose of low-dose aspirin [81 mg, 100 mg, 162 mg, 200 mg,

Others]

Existence of concomitant drug [Yes or No]

(excluding low-dose aspirin)

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup, and chi-square test will be conducted as reference (excluding items falling under the category of multiple counts).

(1) Number of patients with ADRs, etc.

(2) Proportion of patients with ADRs, etc. and its 95% confidence interval (two-sided)

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

#### 4.4.2 Incidence of ADR/infection by sex

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.3 Incidence of ADR/infection by age subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Age (year) [Min<= - <65, 65<= - <75, 75<= - <=Max]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

# 4.4.4 Incidence of ADR/infection by purpose of low-dose aspirin therapy

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Purpose of low-dose aspirin therapy [Angina pectoris, Myocardial

(multiple counts) infarction, Transient ischemic attack

(TIA), Cerebral infarction, Others]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.5 Incidence of ADR/infection by presence/absence of complication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of complication [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

### 4.4.6 Incidence of ADR/infection by presence/absence of renal disease

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of renal disease [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.7 Incidence of ADR/infection by presence/absence of hepatic disease

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of hepatic disease [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

# 4.4.8 Incidence of ADR/infection by BMI subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: BMI ( $kg/m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le - \le Max$ 

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

### 4.4.9 Incidence of ADR/infection by initial daily dose of low-dose aspirin

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Initial daily dose of low-dose [81 mg, 100 mg, 162 mg, 200 mg, Others]

aspirin

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

# 4.4.10 Incidence of ADR/infection by presence/absence of concomitant drug (excluding low-dose aspirin)

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of concomitant drug (excluding low- [Yes or No]

dose aspirin)

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

### 4.4.11 Change of liver function test value

Analysis Safety analysis set

population:

Analysis items: AST (IU/L), ALT (IU/L), γ-GTP (IU/L), ALP (IU/L), Total bilirubin (mg/dL),

LDH (IU/L), Serum gastrin (pg/mL)

Analysis method: Summary statistics will be calculated for the measured values of each

evaluation period [at the start of treatment, at the completion of survey] for the above analysis items. In addition, summary statistics and 95% confidence interval (two-sided) of mean change from the start of treatment with Takecab

Tablets will be calculated.

### 5 Tabulated analysis on efficacy results

# 5.1 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum

Analysis Efficacy analysis set

population:

Analysis items: Development of gastric ulcer, duodenal [Yes or No]

ulcer, or hemorrhagic lesions in stomach or

duodenum

Breakdown (multiple counts)

Development of gastric ulcer [Yes or No]

Development of duodenal ulcer [Yes or No]

Development of hemorrhagic lesions in [Yes or No]

stomach

Development of hemorrhagic lesions in [Yes or No]

duodenum

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

95% confidence interval (two-sided) of proportions of patients who developed

ulcer or hemorrhagic lesions will be calculated.

# 5.2 Development of gastric ulcer, duodenal ulcer, or hemorrhagic lesions in stomach or duodenum (count in each subgroup)

Analysis Efficacy analysis set

population:

Analysis items: Development of gastric ulcer, duodenal [Yes or No]

ulcer, or hemorrhagic lesions in stomach or

duodenum

Breakdown (multiple counts)

Development of gastric ulcer [Yes or No]

Development of duodenal ulcer [Yes or No]

Development of hemorrhagic lesions in [Yes or No]

stomach

Development of hemorrhagic lesions in [Yes or No]

duodenum

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

Existence of *H. pylori* infection [Positive or Negative or Unknown]

BMI (kg/m<sup>2</sup>) [Min<= -<18.5, 18.5<= -<25.0,

 $25.0 \le - \le Max$ 

Initial daily dose of low-dose aspirin [81 mg, 100 mg, 162 mg, 200 mg,

Others]

Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

point estimates and 95% confidence interval (two-sided) of proportions of

patients who developed ulcer or hemorrhagic lesions will be calculated.

# 6 Incidence of ADR/infection in additional pharmacovigilance activities

# 6.1 Incidence of ADR/infection in additional pharmacovigilance activities (Attachment Form 12)

Analysis Safety analysis set

population:

Analysis items: ADRs, etc. falling under the category of safety specification (described as

important identified risks, important potential risks, and important missing

information)

Subgroup items: Seriousness [Serious, Non-serious]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup in accordance with Notes 1 to 4 in Attachment Form 12 included in

PSEHB/PED Notification No. 1128-2 (reexamination notification) dated

November 28, 2017.

(1) Number and proportion of patients with ADRs, etc.

Risk terms and their order of listing will follow those of important identified

risks, important potential risks, and important missing information.

# 7 Outline of patients in postmarketing surveillance, etc.

# 7.1 Outline of patients in postmarketing surveillance, etc. (Attachment Form 16)

Analysis Patients whose survey forms have been collected

population:

Analysis items: Patient number

Name of facility

Sex

Date of birth

Indication (disease code, disease name)

Complication (disease code, disease name)

Route of administration

Maximum dose

Mean dose

Unit

Treatment period

Concomitant drug (drug code, drug name)

Level of effect

ADR (disease code, disease name, outcome)

Survey form No.

Withdrawal

Analysis method: A list will be prepared for the above analysis items in accordance with Notes 1 to

3 in Attachment Form 16 included in PSEHB/PED Notification No. 1128-2

(reexamination notification) dated November 28, 2017.

**Revision history (version control)** 

| Version | Date | Person who prepared/revised this document | Comment |
|---|---|---|---|
| Version 1 | 2019.8.7 | PPD | Preparation of Version 1 |